CLINICAL TRIAL: NCT05010317
Title: Acceptability, Feasibility and Effectiveness of a Mindfulness Based Intervention to Promote Adherence to Antiretroviral Therapy Among Adolescents in Kampala.
Brief Title: Mindfulness and Acceptance Based Therapy for Adolescents Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Collaborators: Makerere University (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D43TW011304 (NIH); D43TW011304 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2021-08-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-05

CONDITIONS: Medication Adherence; Adjustment Reaction With Anxiety and Depression; Mental Health Issue
MeSH Terms: conditions — Medication Adherence; Depression | interventions — Mindfulness; Acceptance and Commitment Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: One group of adolescents (treatment group), will be exposed to a mindfulness and acceptance based psychotherapy on top of usual clinic care services, while the other group will keep receiving usual clinic care. Then comparison will be made at post intervention on experiences of depression, stigma, anxiety, psychological flexibility and then self-reported medical adherence at post intervention between the two groups, adjusting for baseline measures.
Masking Description: This will be an open label randomized study because the staff will be involved in the care of the participants, assessment of the outcome and the nature of the psychosocial interventions to be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving the mindfulness and acceptance intervention (Experimental): This group will under go four sessions of the mindfulness and acceptance based therapy. These sessions will be delivered in four weeks, utilizing 2 hours every week. This will be in addition to the standard of care (clinic based counselling).
  Interventions: Behavioral: Mindfulness and acceptance based therapy; Behavioral: Standard of care
- Control group (Active Comparator): This group will continue receiving the usual clinic based care (counselling) only.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Mindfulness and acceptance based therapy — This is a behavioral intervention that is aimed at building psychological flexibility among adolescents. It involves careful use of language, metaphors, experiential learning and mindfulness to develop skills that support values guided living. Participants learn to relate with their inner thoughts, feelings and urges in an open and elaborative way as conscious human beings and make choices that improve their lives even in the presence of such difficult experiences.
  Other Names: Acceptance and commitment therapy; Discoverer, Noticer, Advisor-Values
  Arms: Group receiving the mindfulness and acceptance intervention
Behavioral: Standard of care — Usual clinic based counselling offered as routine care to adolescents

SUMMARY:
Adolescents represent a growing share of people living with HIV in sub-Saharan Africa (SSA), yet show poor adherence to medication and viral suppression (VS) compared to adults. Investigators postulate that to achieve optimal adherence, support interventions that resonate with life-stages changes in adolescence need to be tested and promoted. Mindfulness and acceptance based interventions are slowly gaining traction as appropriate for adolescents.

The study proposes to explore acceptability of an adapted mindfulness and acceptance-based psychosocial intervention (acceptance and commitment therapy: Discoverer, Noticer, Advisor-values model-ACT-DNA-v), among providers (health care practitioners -HCPs) and users (adolescents living with HIV/AIDS-ALWHA). Further, it endeavors to measure feasibility and effectiveness of ACT-DNA-v in reducing psychological barriers to adherence among ALWHAs. The study is to be conducted at two public health centers in Kampala-Uganda. The study design is exploratory sequential mixed-methods; where qualitative data is to be used to explore acceptance of ACT-DNA-v, while quantitative data will be used to measure feasibility of the intervention and its effectiveness in reducing psychosocial barriers to adherence. Qualitative exploratory methods will guide exploration of acceptability of ACT-DNA-v among users and providers; collecting data with a semi-structured interview on domains of inquiry including; understanding, satisfaction, intention to use and perceived appropriateness of ACT-DNA-v. A randomized control trial with quantitative surveys at baseline, post-intervention and follow-up will used to measure the effects of the intervention on process and clinical outcomes among ALWHA. Thematic data analysis will be used to analyze qualitative data, while T-test, Wilcoxon rank sum test, Fisher's exact and Chi-square tests respectively will be used to ascertain average mean differences between the ACT group and the control group on the outcome parameters.

DETAILED DESCRIPTION:
Background The success of antiretroviral therapy (ART) is highly dependent on adherence and persistent care engagement. However, despite efforts to improve sustained ART use among adolescents, non-adherence persists. Studies using medication possession ratios and clinical counts have found adherence to ART among adults to be at 72% compared to 68% among young people, furthermore, statistics on VL measures in 2017 show that 74.2% of adults above 50 years had achieved viral load suppression compared to 39.6% of adolescents. Additionally, almost 50% of HIV cases in Uganda are among young people. Poor adherence among ALWHA undermines the HIV care cascade and efforts to end the AIDS epidemic by 2030. As a consequence, young people are the only group in Uganda among whom HIV mortality is increasing. The unique developmental changes at the onset of adolescence have been cited as main factors influencing psychosocial pathways into health, resulting in psychopathological barriers to medication adherence among ALWHA. Developmentally appropriate psychosocial interventions need to be added into adolescents' HIV care. However, to date, psychosocial support interventions targeted for the unique developmental changes in adolescence remain limited. Most interventions in use with young people are developed for adult populations, despite adult-focused interventions being shown to have limited effectiveness among young people. Besides, some interventions like short message services are expensive and difficult to sustain, while others lack a clear mechanism of change for replication.

Mindfulness and acceptance based interventions, specifically ACT-DNA-v, are developmentally appropriate for adolescents because they are designed to promote emotion regulation and values consistent living, counteracting the imbalance created by developmental changes amidst undeveloped executive functions such as judgment. Besides, ACT-DNA-v relies on use of art and metaphors which serve as aids to symbolic reasoning (a change instigated by adolescence). The intervention is also centered around values and adolescence is a stage of establishing identity. Finally, ACT-DNA-V has a proper mechanism of change called psychological flexibility, thus, it can easily be replicated. However, while mindfulness and acceptance based interventions have been found to be effective in improving mental health of adolescents in the developed world, they have not been tested in resource limited settings, with adolescents living with HIV and for outcomes beyond mental health. Thus, this study set out to adapt ACT-DNA-v for use in a resource limited setting, explore its acceptability among users (ALWHAs) and providers (HCPs), measure its feasibility when used with adolescents and evaluate its impact on reducing psychosocial barriers to adherence, improve self-reported adherence and reducing viral load.

Study Objectives The study aims to achieve the following objectives;

.To adapt and explore acceptability of ACT-DNA-v among users (ALWHA) and providers (HCPs).

.To measure feasibility of the adapted ACT-DNA-v for use with ALWHA.

.To examine the impact of ACT-DNA-v on reducing proximal psychosocial barriers to medication adherence (depression, anxiety and stigma) among ALWHA.

.To measure effectiveness of a mindfulness based intervention (ACT-DNA-v) on self-reported adherence among ALWHA in Kampala, and ascertain its impact on viral load reduction via analysis of data from medical records

Hypothesis .Participants receiving the ACT-DNA-v intervention will report a significant reduction in depression, anxiety & stigma at four months' follow-up as compared to participants in the control group.

.Participants receiving the ACT-DNA-v intervention will have significantly higher levels of reported ART adherence and lowered viral load at four months' follow-up compared to participants not receiving this intervention.

Methods Overall design To achieve the study goals, a mixed methods design will be used, specifically exploratory sequential. The mixing is intended for purposes of expansion (where qualitative data will explore acceptability of the mindfulness based intervention and quantitative data measures if the accepted intervention is effective). This will improve the usefulness of the findings, (qualitative data evaluating the process while quantitative data evaluate the outcomes). The study will involve two sub-studies; formative/qualitative study and intervention/quantitative study.

ELIGIBILITY:
Inclusion Criteria:

* Participant should be 15-19 years of age.
* Diagnosed HIV positive.
* Attending care at the two study sites (Kisenyi and Kitebi) for the last 6 months.
* On first or second line of treatment.
* Can speak/understand Luganda or English.
* Willing to provide informed consent/assent.
* All records will be confirmed via clinic medical charts.

Exclusion Criteria:

* A participant plan to move out of the catchment area within six months.
* Participant is participating in another study related to HIV and care improvement.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in levels of Depression; measured by Beck's Depression Inventory-ii | pre-intervention and at four weeks post intervention assessment
  The outcome measure will be; number of participants in a given study group reporting change from baseline depression levels at post intervention and after three months follow-up. The change will be assessed by Beck's depression inventory-ii. According to the BDI-ii, scores in the range of 0-13 represent minimal depression, 14-19 mild depression, 20-28 moderate, while 29-63 severe depression.
Change in Health related anxiety; measured by the short health anxiety inventory | At pre-intervention and at four weeks post intervention assessment
  The outcome measure will be number of participants in a given study arm reporting change from baseline health anxiety at post intervention and at three months follow-up. According to the SHAI, 40.5 is the cut-off score separating clinical and non-clinical health related anxiety.
Change in AIDS related Internalized stigma; measured by Internalized AIDS related stigma scale (IARSS-6) | At pre-intervention and at four weeks post intervention assessment
  After dichotomizing the IARSS-6 at median value (0-2 & 3-6), two categories will be created. Category 1 is in the 0-2 range (representing low-moderate stigma) while category 2 is the 3-6 range (representing higher experience of stigma). The measure will then be; the number of participants in a given study arm reporting change from baseline AIDS related stigma at post intervention and at three months follow-up as assessed by the internalized AIDS related stigma scale.

SECONDARY OUTCOMES:
Self-reported medication adherence; measured by the Morisky Medication Adherence scale-MMAS-8. | At three months
  The 3 categorical Likert Scale is low adherence = <6, medium adherence = 6-<8 and high adherence is = 8.
Viral load | At three months
  This measure will be based on clinic records. Viral load measures (copies/milliliter of blood) for each participant in both groups will be recorded at baseline and at follow-up. A comparison will be made to detect if there is a difference at time points and across groups.

OTHER OUTCOMES:
Psychological flexibility; measured by the Avoidance and Fusion Questionnaire for youths (AFQ-Y8). | At three months
  This is a process measure and mechanism of change. AFQ-Y8 measures cognitive fusion and experiential avoidance as impediments to attaining Psychological Flexibility. Scores of the AFQ-Y8 range from 0-24, with higher scores indicating higher levels of psychological inflexibility. The outcome measure for Psychological flexibility will be the number of participants in a given study arm reporting change from baseline psychological inflexibility at post intervention and at three months follow-up as assessed by the AFQ-Y8.

CONTACTS AND LOCATIONS:
Overall Officials: Moses R Kamya, Study Chair — IDRC
Locations (2):
- Uganda (2):
  - Kisenyi Health center iv, Kampala, Central Region
  - Kitebi health center iii, Kampala, Non-US/Non-Canadian

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessed through a public repository or upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available effective 1st June 2023. It will remain available for one year
Access Criteria: through clinicaltrials.gov

REFERENCES:
- [Background] Soomro N, Fitzgerald G, Seeley J, Schatz E, Nachega JB, Negin J. Comparison of Antiretroviral Therapy Adherence Among HIV-Infected Older Adults with Younger Adults in Africa: Systematic Review and Meta-analysis. AIDS Behav. 2019 Feb;23(2):445-458. doi: 10.1007/s10461-018-2196-0. PMID 29971732
- [Background] Burckhardt R, Manicavasagar V, Batterham PJ, Hadzi-Pavlovic D, Shand F. Acceptance and commitment therapy universal prevention program for adolescents: a feasibility study. Child Adolesc Psychiatry Ment Health. 2017 May 25;11:27. doi: 10.1186/s13034-017-0164-5. eCollection 2017. PMID 28559924
- [Background] Casale M, Carlqvist A, Cluver L. Recent Interventions to Improve Retention in HIV Care and Adherence to Antiretroviral Treatment Among Adolescents and Youth: A Systematic Review. AIDS Patient Care STDS. 2019 Jun;33(6):237-252. doi: 10.1089/apc.2018.0320. PMID 31166783
- [Background] Vreeman RC, McCoy BM, Lee S. Mental health challenges among adolescents living with HIV. J Int AIDS Soc. 2017 May 16;20(Suppl 3):21497. doi: 10.7448/IAS.20.4.21497. PMID 28530045
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Kalichman SC, Simbayi LC, Cloete A, Mthembu PP, Mkhonta RN, Ginindza T. Measuring AIDS stigmas in people living with HIV/AIDS: the Internalized AIDS-Related Stigma Scale. AIDS Care. 2009 Jan;21(1):87-93. doi: 10.1080/09540120802032627. PMID 19085224
- [Background] Moon SJ, Lee WY, Hwang JS, Hong YP, Morisky DE. Accuracy of a screening tool for medication adherence: A systematic review and meta-analysis of the Morisky Medication Adherence Scale-8. PLoS One. 2017 Nov 2;12(11):e0187139. doi: 10.1371/journal.pone.0187139. eCollection 2017. PMID 29095870
- [Background] Greco LA, Lambert W, Baer RA. Psychological inflexibility in childhood and adolescence: development and evaluation of the Avoidance and Fusion Questionnaire for Youth. Psychol Assess. 2008 Jun;20(2):93-102. doi: 10.1037/1040-3590.20.2.93. PMID 18557686
- [Background] Abramowitz JS, Deacon BJ, Valentiner DP. The Short Health Anxiety Inventory: Psychometric Properties and Construct Validity in a Non-clinical Sample. Cognit Ther Res. 2007;31(6):871-883. doi: 10.1007/s10608-006-9058-1. Epub 2007 Feb 15. PMID 32214558
- [Derived] Musanje K, Kasujja R, Camlin CS, Hooper N, Hope-Bell J, Sinclair DL, Kibanja GM, Mpirirwe R, Kalyango JN, Kamya MR. Effectiveness of a mindfulness and acceptance-based intervention for improving the mental health of adolescents with HIV in Uganda: An open-label trial. PLoS One. 2024 May 9;19(5):e0301988. doi: 10.1371/journal.pone.0301988. eCollection 2024. PMID 38722926
- See also: UPHIA Uganda factsheet — https://www.afro.who.int
- See also: UNAIDS report on the global AIDS epidemic 2020 — http://www.unaids.org